CLINICAL TRIAL: NCT03732157
Title: Feasibility of Parathyroidectomy With Exploration of 4 Parathyroid Glands in Outpatients, for Treatment of Primary Hyperparathyroidism
Brief Title: Feasibility of Parathyroidectomy With Exploration of 4 Parathyroid Glands in Outpatients
Acronym: PARAMBU
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K180301J
Record Dates: First submitted 2018-09-18; First posted 2018-11-06 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-09

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; Parathyroidectomy; Outpatient management
MeSH Terms: conditions — Hyperparathyroidism, Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- outpatient management of parathyroidectomy
  Interventions: Procedure: outpatient management of parathyroidectomy
- conventional management of parathyroidectomy
  Interventions: Procedure: conventional management of parathyroidectomy

INTERVENTIONS:
Procedure: outpatient management of parathyroidectomy — The patient is discharged from hospital the same day of the parathyroidectomy intervention instead of conventional management (stay overnight in hospital)
  Groups: outpatient management of parathyroidectomy
Procedure: conventional management of parathyroidectomy — The patient stays overnight in hospital after intervention
  Groups: conventional management of parathyroidectomy

SUMMARY:
The development of outpatient surgery has become a national priority, with the objective of an ambulatory surgery rate of around 50% in 2016, whereas this rate reached only 37.7% in 2010.

In the context of the management of primary hyperparathyroidism, there are two possible approaches. The first, which is commonly performed on an outpatient basis, consists in approaching only the pathological gland, if it was first identified by scintigraphy and ultrasound (which is the case in one patient in two), without exploring the others parathyroid glands.

The reference technique consists in exploring the 4 parathyroid sites by transverse cervicotomy. Although more invasive, it minimizes the risk of failure due to the lack of knowledge of multi-glandular forms of the disease (15 to 20%), whose preoperative diagnosis is difficult. This reference technique is poorly performed on an outpatient basis while it lends itself to this type of management because of the superficial character of the operative site, a short operating time, moderate postoperative pain, rapid return oral nutrition and exceptional and early serious complications (delay <24 h for cervical hematoma, <24 h for hypocalcemia and immediate diagnosis of recurrent palsy).

In this study, the investigators hypothesize that parathyroidectomy with 4-gland parathyroid exploration is feasible by ensuring patient safety. The investigators also believe that outpatient management will not lead to any difference after 3-month surgery, but will reduce hospitalization costs while increasing patient satisfaction with conventional care. To do so, the investigators carried out an observational cohort study of patients with an indication of parathyroidectomy wo will undergo outpatient management or conventional management (stay overnight in hospital) to inform all of these data.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Diagnosis of primary hyperparathyroidism (inappropriate parathyroid hormone secretion compared with calcemia)
* Surgical indication of parathyroidectomy with possible management outpatient or conventional hospitalization (choice of mode of care by the surgeon, after consultation with the patient)

Exclusion Criteria:

* Non-eligibility for outpatient surgery for general medical reasons (ASA score), determined during the consultation of preoperative anesthesia
* Preoperative hypercalcemia> 3 mmol / L (due to the high risk of postoperative hypocalcemia)
* History of cervicotomy for thyroidectomy or failure of parathyroid surgery
* Treatment of primary hyperparathyroidism with elective surgical approach
* Person under guardianship and curatorship

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients with primary hyperparathyroidism
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of conversion or readmission to conventional hospitalization | within 8 days postoperatively
  The primary endpoint will be assessed for patients receiving outpatient management. Proportion of patients who could not discharged from hospital the same day of surgery as originally scheduled or being readmitted to conventional hospitalization within 8 days post operatively.

SECONDARY OUTCOMES:
Postoperative pain evaluated using visual analogue scale (VAS) | at day 0 post operatively
  Pain will be evaluated using visual analogue scale (VAS) . VAS score ranges from 0 to 10. A high VAS score represents a high level of pain while a low VAS score represents a low level of pain.
Postoperative pain evaluated using visual analogue scale (VAS) | at day 1 post operatively
  Pain will be evaluated using visual analogue scale (VAS) . VAS score ranges from 0 to 10. A high VAS score represents a high level of pain while a low VAS score represents a low level of pain.
Postoperative pain evaluated using visual analogue scale (VAS) | at day 8 post operatively
  Pain will be evaluated using visual analogue scale (VAS) . VAS score ranges from 0 to 10. A high VAS score represents a high level of pain while a low VAS score represents a low level of pain.
Proportion of patients with breathing difficulty. | at day 1 post operatively
  Dyspnea will be evaluated using the New York Heart Association (NYHA) Functional Classification. The stage of dyspnea is classified in four categories based on how much patients are limited during physical activity. Breathing difficulty will be defined by a stage of 3 on the NYHA scale.
Proportion of patients with breathing difficulty. | at day 8 post operatively
  Dyspnea will be evaluated using the New York Heart Association (NYHA) Functional Classification. The stage of dyspnea is classified in four categories based on how much patients are limited during physical activity. Breathing difficulty will be defined by a stage of 3 on the NYHA scale.
Proportion of patients with compressive cervical hematoma | at day 0 post operatively
  clinical evaluation based on the occurrence of a cervical collection that can obstruct the upper aero-digestive tract (NYHA scale dyspnea)
Proportion of patients with compressive cervical hematoma | at day 1 post operatively
  clinical evaluation based on the occurrence of a cervical collection that can obstruct the upper aero-digestive tract (NYHA scale dyspnea)
Proportion of patients with compressive cervical hematoma | at day 8 post operatively
  clinical evaluation based on the occurrence of a cervical collection that can obstruct the upper aero-digestive tract (NYHA scale dyspnea)
Proportion of patients with hypocalcemia | at day 1 post operatively
  Hypocalcemia will be defined as calcemia lower than 2 mmol/L or 80 mg/L
Proportion of patients with hypocalcemia | at 3 months post operatively
  Hypocalcemia will be defined as calcemia lower than 2 mmol/L or 80 mg/L
Proportion of patients with recurrent nerve paralysis | at day 0 post operatively
  Clinical evaluation based on the occurrence of voice modification with swallowing disorder
Proportion of patients with recurrent nerve paralysis | at day 1 post operatively
  Clinical evaluation based on the occurrence of voice modification with swallowing disorder
Proportion of patients with recurrent nerve paralysis | at day 8 post operatively
  Clinical evaluation based on the occurrence of voice modification with swallowing disorder
Patients' satisfaction regarding his/her care evaluated using visual analogue scale (VAS) | at day 0 post operatively
  Patients' satisfaction evaluated using visual analogue scale (VAS). VAS score ranges from 0 to 10. A high VAS score represents a high level of satisfaction while a low VAS score represents a low level of satisfaction.
Patients' satisfaction regarding his/her care evaluated using visual analogue scale (VAS) | at day 1 post operatively
  Patients' satisfaction evaluated using visual analogue scale (VAS). VAS score ranges from 0 to 10. A high VAS score represents a high level of satisfaction while a low VAS score represents a low level of satisfaction.
Patients' satisfaction regarding his/her care evaluated using visual analogue scale (VAS) | at 3 months post operatively
  Patients' satisfaction evaluated using visual analogue scale (VAS). VAS score ranges from 0 to 10. A high VAS score represents a high level of satisfaction while a low VAS score represents a low level of satisfaction.
Total cost of mode of care | at 3 months post operatively
  Total cost of hospital surgery stay and hospital readmission at 3 months

IPD SHARING:
Plan to Share IPD: Undecided